CLINICAL TRIAL: NCT02809261
Title: The Long-term Effect of Perineural Injection Therapy in Patients With Carpal Tunnel
Brief Title: The Effect of Perineural Injection Therapy in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending physician of physical medicine and rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB No: 2-105-05-033
Record Dates: First submitted 2016-06-10; First posted 2016-06-22 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Perineural injection; Dextrose
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perineural injection with 5% dextrose (Experimental): Ultrasound-guided perineural injection with 5% Dextrose (3cc) between proximal carpal tunnel and median nerve.
  Interventions: Procedure: Ultrasound-guided perineural injection with 5% dextrose; Drug: 5% Dextrose
- Perineural injection with normal saline (Placebo Comparator): Ultrasound-guided perineural injection with normal saline (3cc) between proximal carpal tunnel and median nerve.
  Interventions: Procedure: Ultrasound-guided perineural injection with normal saline; Drug: Normal Saline

INTERVENTIONS:
Procedure: Ultrasound-guided perineural injection with 5% dextrose — Ultrasound-guided perineural injection with 5% dextrose (3cc) between proximal carpal tunnel and surrounding median nerve with hydrodissection.
  Arms: Perineural injection with 5% dextrose
Procedure: Ultrasound-guided perineural injection with normal saline — Ultrasound-guided perineural injection with normal saline (3cc) between proximal carpal tunnel and surrounding median nerve with hydrodissection.
  Arms: Perineural injection with normal saline
Drug: Normal Saline — Normal saline is safe for perineural injection.
  Arms: Perineural injection with normal saline
Drug: 5% Dextrose — 5% Dextrose could decrease the release of CGRP and substance P to reduce the nerve inflamation.
  Arms: Perineural injection with 5% dextrose

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. Although many conservative managements of CTS, the effectiveness of these methods is insignificant or only persist for a short duration. Recently, the ultrasound-guided perineural injection with 5% dextrose was widely used for entrapment neuropathy with positive benefit. However, current studies have not entirely proved the effects of perineural injection on peripheral neuropathy because these studies enrolled small number of patients and lacked controlled design. The investigators design a randomized, double-blind, controlled trail to assess the effect after ultrasound-guided perineural injection with 5% dextrose in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically diagnosed with CTS were randomized into intervention and control group. Participants in intervention group received one-session ultrasound-guided perineural injection with 5% dextrose and control group received one-session ultrasound-guided perineural injection with normal saline. No additional treatment after injection through the study period. The primary outcome is visual analog scale (VAS) and secondary outcomes include Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd, 4th, 8th, 12th, 16th and 24th week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-85 year-old.
* Diagnosis was confirmed using an electrophysiological study and ultrasonography

Exclusion Criteria:

Cancer

* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the symptoms and functional status before treatment and multiple time frame after treatment
Change from baseline in cross-sectional area of the median nerve on 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment. | Pre-treatment, 2nd, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Mulvaney SW. Ultrasound-guided percutaneous neuroplasty of the lateral femoral cutaneous nerve for the treatment of meralgia paresthetica: a case report and description of a new ultrasound-guided technique. Curr Sports Med Rep. 2011 Mar-Apr;10(2):99-104. doi: 10.1249/JSR.0b013e3182110096. PMID 21623291
- [Result] Tsui BC, Wagner A, Finucane B. Electrophysiologic effect of injectates on peripheral nerve stimulation. Reg Anesth Pain Med. 2004 May-Jun;29(3):189-93. doi: 10.1016/j.rapm.2004.02.002. PMID 15138901
- [Result] Tsui BCH, Kropelin B. The electrophysiological effect of dextrose 5% in water on single-shot peripheral nerve stimulation. Anesth Analg. 2005 Jun;100(6):1837-1839. doi: 10.1213/01.ANE.0000153020.84780.A5. PMID 15920223
- [Derived] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254